CLINICAL TRIAL: NCT07299604
Title: Effect of Chronic Exercise on Human Thermogenic Adipose Tissue & Elucidation of Mechanisms
Acronym: ExBat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: German Research Foundation (Other); University Hospital, Bonn (Other); Helmholtz Center Munich (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-ExBat; TRR333 (Other Grant/Funding Number: German Research Fondation, SFB)
Record Dates: First submitted 2025-11-14; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Endurance Training; No Training
Keywords: brown adipose tissue; activation; endurance training; oxygen consumption
MeSH Terms: interventions — Endurance Training

STUDY DESIGN:
Intervention Model Description: The investigators will recruit 24 participants, who will be randomised into two arms: 1) 6 weeks of individualised/supervised endurance training; 2) a control group without any additional training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endurance training (Experimental): The participants fulfill an individualized and supervised training. The 6 weelk training period consits of three training sessions per week.
  Interventions: Behavioral: Endurance Training
- Control group (No Intervention): In parallel to the intervention group the control group only fulfill the inclusion measures and the follow-up measusres without any additional training. They will be advised to keep constant there normal physical activity, which has to be documented in dairy book.

INTERVENTIONS:
Behavioral: Endurance Training — 6 weeks of endurance training, 3time per week
  Arms: Endurance training

SUMMARY:
Physical exercise can stimulate heat production in our bodies. This is healthy because it burns sugar and fat. Heat production is influenced, among other things, by what is known as 'brown or beige adipose tissue', which is capable of producing heat in our bodies. However, everyone reacts differently to physical exercise. In addition, different types of exercise can influence heat production. That is why the investigators want to use this study to investigate why different people show different reactions in brown and beige adipose tissue. This is important for our metabolism and our health.

The study will last approximately 6 weeks. The participants are healthy individuals who are participating in the study. The test subjects will be divided into two groups by drawing lots, so that there are equal numbers of men and women in each group.

One group will complete a 6-week endurance training programme. The other group (control) will not do any additional training and will serve as a control group. However, the accompanying examinations will be the same for both groups. By comparing the two groups, the investigators will be able to see whether training has a better effect on heat production and thus health.

As part of this study, the investigators want to investigate how 6 weeks of endurance training affects the function of brown and beige adipose tissue. To do this, the investigators will take some blood and adipose tissue samples before and after the training period.

DETAILED DESCRIPTION:
In order to investigate the regulation of thermogenic adipose tissue by physical exercise and other stimuli without the need for biopsies, the investigators have developed a cell assay that allows to investigate the effect of sera taken before or after physical exertion, e.g. on the expression of the heat-generating UCP1 protein. Experiments using this test have shown that exercise-conditioned serum stimulates UCP1 expression on average compared to resting serum. However, the increase in UCP1 expression in athletes is more than twice as high and there are large inter-individual variations, i.e. non-responders, average responders and 'super responders'. This implies that some subjects secrete serum factors during exercise that can activate thermogenesis in adipose tissue.

It is also known that immune cells have an effect on adipose tissue and may also be involved in crosstalk. Therefore, the aim here is to investigate the reactivity of immune cells using single-cell mRNA sequencing. This analysis may provide further insight into immune responses, including in relation to obesity.

Using this methodology, the investigators now want to investigate how acute physical exercise 6-week training intervention (endurance training) influence the thermogenic adipose tissue, metabolism and energy expenditure of the participants.

The investigators have three specific objectives:

1. The investigators will analyse how serum taken before or after training affects the expression of the heat-generating UCP1 protein in human adipocytes in cell culture. The investigators will also measure oxygen consumption/energy expenditure during cold stimulation and correlate these measurements with those obtained in adipocyte cell cultures. Furthermore, the investigators will quantify mRNA expression in isolated immune cells (peripheral mononuclear cells and granulocytes).
2. The investigators will use the sera, cells and biopsy samples obtained to analyse the mechanisms of white/beige adipose tissue regulation in cooperation with the project consortium. One focus will be on miRNAs in exosomes, which have been identified as biomarkers for thermogenesis. In addition, the investigators will add thermogenic super-responder sera and non-thermogenic non-responder sera to human adipocytes in cell culture and perform a phosphoproteomics analysis. Based on this analysis, the investigators will then attempt to identify the factors that activate thermogenesis.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-25
* male/female
* less than 3 hours/week of regular training
* must be able to perform performance analysis and endurance training by cycling
* must be able to do six weeks of training

Exclusion Criteria:

* cardiovascular, pulmonary, neoplastic, orthopaedic, metabolic, or chronic diseases
* problems that preclude performance testing or endurance testing
* pregnancy (only female)
* regular medication
* smoking
* dependency relationship with the TUM Professorship of Exercise Biology

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
UCP-1 gene expression in cultured adipocytes treated with conditioned human sera | Serum samples will be collected at baseline and after six week of endurance training or six week of control period. Cell culture experiments will start when the last participant completed the study.
  The investigators collect human serum samples before/after training/control period and before/after cold exposure and exercise testing. Human adipose tissue cells will be treated with the conditioned serum samples of the training and control groups. The primary outcome measure is the change of mRNA expression of UCP-1 in adipose tissue cells by PCR.

SECONDARY OUTCOMES:
Energy expenditure in reaction to cold exposure | Cold exposure will be done before and after the training or control period of six weeks.
  The investigators will measure oxygen consumption during a one-hour period of cold exposure.
Physical performance analysis (oxygen consumption in ml/kg body weight) | Physical performance analysis will be done before and after the training or control period of six weeks.
  Before and after the training or control intervention, participants undergo cardio-pulmonary exercise testing to assess their physical performance. The investigators will measure oxygen consumption during an incremental cycling test.
Physical performance analysis (heart rate in bpm) | Physical performance analysis will be done before and after the training or control period of six weeks.
  Before and after the training or control intervention, participants undergo cardio-pulmonary exercise testing to assess their physical performance. The investigators will measure heart rate during an incremental cycling test.
Physical performance analysis (blood lactate in mmol/L) | Physical performance analysis will be done before and after the training or control period of six weeks.
  Before and after the training or control intervention, participants undergo cardio-pulmonary exercise testing to assess their physical performance. The investigators will measure lactate production after each stage during an incremental cycling test.
Physical performance analysis (power output in W) | Physical performance analysis will be done before and after the training or control period of six weeks.
  Before and after the training or control intervention, participants undergo cardio-pulmonary exercise testing to assess their physical performance. The investigators will measure maximal power output on the bicycle ergometer during an incremental step test until voluntary maximal exhaustion.
Supraclavicular skin temperature in response to cold exposure | Cold exposure will be done before and after the training or control period of six weeks.
  The investigators will measure supraclavicular skin temperature during a one-hour period of cold exposure.

OTHER OUTCOMES:
exomiRs screening by PCR/sequencing | Serum samples will be collected at baseline and after six week of endurance training or six week of control period. Cell culture experiments will start when the last participant.
  ExomiRs will be obtained from blood sera as well as cell culture supernatants by differential ultracentrifugation. Subsequently, the microRNAs are then isolated from the exosomes and quantified by PCR/sequencing.
Metabolomics screening (relative quantities) | Plasma samples will be collected at baseline and after six week of endurance training or six week of control period.
  To expand the mechanistic investigations, sera/cell culture supernatants will be screened for changes in metabolites. For this purpose, the samples are evaluated using untargeted mass spectrometry.
Proteomics screening (relative quantities) | Plasma samples will be collected at baseline and after six week of endurance training or six week of control period.
  To expand the mechanistic investigations, sera/cell culture supernatants will be screened for changes in protein quantities. For this purpose, the samples are evaluated using untargeted mass spectrometry.
UCP-1 gene expression in human adipose tissue biopsies | Adipose tissue biopsies will be collected at baseline and after six week of endurance training or six week of control period. Analysis of samples will start when the last participant completed the study.
  The investigators collect human adipose tissue biopsy samples before/after training/control period. The outcome measure is the change of mRNA expression of UCP-1 in the adipose tissue biopsies by PCR.
Single-cell sequencing analysis of isolated immune cells after acute endurance exercise | Immune cells will be isolated before and after acute endurance exercise from venous blood of 8 untrained participants (4 women and 4 men).
  Immune cells will be isolated from peripheral blood mononuclear cells for single-cell sequencing analysis. Immune cell population and respective gene expression will be compared between resting and exercised conditions among both women and men.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Braunsperger, PhD candidate, Study Chair — Technical University Munich, Professorship of Exercise Biology, Am Olympacampus 11, 80809 Munich
Locations (1):
- University Munich, Professorship of Exercise Biolog, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project website — https://www.hs.mh.tum.de/exercisebiology/forschung-publikationen/exbat-sfb/